CLINICAL TRIAL: NCT00082940
Title: A Phase II Study of ONTAK® (Denileukin Diftitox, DABIL-2) in Patients With Fludarabine-Refractory B-Cell Chronic Lymphocytic Leukemia
Brief Title: Denileukin Diftitox in Treating Patients With Fludarabine-Refractory B-Cell Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CCCWFU-27102; CDR0000361734 (Registry Identifier: PDQ (Physician Data Query)); CCCWFU-BG02-331; LIGAND-CCCWFU-27102
Record Dates: First submitted 2004-05-14; First posted 2004-05-19 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2013-06

CONDITIONS: Leukemia
Keywords: B-cell chronic lymphocytic leukemia; refractory chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — denileukin diftitox

INTERVENTIONS:
Biological: denileukin diftitox

SUMMARY:
RATIONALE: Biological therapies, such as denileukin diftitox, may interfere with the growth of cancer cells and slow the growth of chronic lymphocytic leukemia.

PURPOSE: This phase II trial is studying how well denileukin diftitox works in treating patients with fludarabine-refractory B-cell chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the complete and partial response rate in patients with fludarabine-refractory B-cell chronic lymphocytic leukemia treated with denileukin diftitox.

Secondary

* Determine the toxicity profile of this drug in these patients.
* Determine the response rate in patients (regardless of CD25 receptor density) treated with this drug.
* Determine the progression-free survival and overall survival of patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive denileukin diftitox IV over 1 hour on days 1-5. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.

Patients achieving a complete response after 8 courses proceed to follow-up. Patients achieving a partial response or stable disease after 8 courses may continue treatment at the discretion of the investigator.

Patients are followed every 3 months for 1 year and then annually until relapse.

PROJECTED ACCRUAL: A total of 12-44 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of B-cell chronic lymphocytic leukemia (CLL) meeting the following criteria at any time during the course of disease (e.g., at initial diagnosis or relapse):

  * Absolute lymphocytosis > 5,000/mm^3
  * Lymphocytes must appear mature with < 55% prolymphocytes
  * More than 30% of all nucleated cells are lymphoid on bone marrow aspirate smear
  * Lymphoid infiltrates compatible with bone marrow involvement by CLL on core bone marrow biopsy
  * Predominant B-cell monoclonal population of cells share the B-cell marker (CD19) with the CD5 antigen in the absence of other pan-T-cell markers by lymphocyte immunophenotyping
* High-risk disease OR intermediate-risk disease

  * Patients in the intermediate-risk group must have evidence of active disease as demonstrated by at least 1 of the following criteria:

    * Massive or progressive splenomegaly and/or adenopathy
    * Weight loss > 10% within the past 6 months
    * Common toxicity grade 2-4 fatigue
    * Fevers > 100.5°F OR night sweats for more than 2 weeks without evidence of infection
    * Progressive lymphocytosis with an increase of > 50% over a 2-month period or an anticipated doubling time of < 6 months
* Failed at least 1 prior fludarabine regimen, as defined by 1 of the following criteria:

  * Refractory or intolerant to fludarabine
  * Relapsed within 6 months after completion of fludarabine
* No CNS leukemia
* No mantle cell lymphoma in leukemic phase

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-2

Life expectancy

* More than 2 months

Hematopoietic

* Absolute neutrophil count ≥ 1,000/mm^3
* Platelet count ≥ 50,000/mm^3
* Hemoglobin ≥ 8 g/dL (transfusion allowed)

Hepatic

* Albumin ≥ 3 g/dL
* AST and ALT ≤ 2.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* No hepatitis B or C infection

Renal

* Creatinine ≤ 1.5 mg/dL OR
* Creatinine clearance ≥ 40 mL/min

Cardiovascular

* LVEF ≥ 40%

Other

* No uncontrolled infection
* No other concurrent serious illness
* No HIV infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use two effective methods of contraception (one must be non-hormonal) during and for at least 1 month after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Prior denileukin diftitox allowed

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* No concurrent corticosteroids as anti-emetics

Radiotherapy

* No concurrent radiotherapy

Surgery

* Not specified

Other

* At least 28 days since prior anticancer therapy and recovered
* No other concurrent antineoplastic drugs

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-08; Primary Completion 2005-01 (Actual); Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur E. Frankel, MD, Study Chair — Wake Forest University Health Sciences
Locations (11):
- United States (11):
  - St. Joseph Hospital Regional Cancer Center - Orange, Orange, California
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Medical Center Vincennes, Vincennes, Indiana
  - Cancer Care Specialists, Houma, Louisiana
  - Feist-Weiller Cancer Center at Louisiana State University Health Sciences, Shreveport, Louisiana
  - Josephine Ford Cancer Center at Henry Ford Health System, Detroit, Michigan
  - Southeastern Medical Oncology Center, Goldsboro, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Chattanooga Oncology and Hematology Associates, Chattanooga, Tennessee
  - Southwest Regional Cancer Center - Central, Austin, Texas

REFERENCES:
- [Result] Frankel AE, Surendranathan A, Black JH, White A, Ganjoo K, Cripe LD. Phase II clinical studies of denileukin diftitox diphtheria toxin fusion protein in patients with previously treated chronic lymphocytic leukemia. Cancer. 2006 May 15;106(10):2158-64. doi: 10.1002/cncr.21851. PMID 16586495